CLINICAL TRIAL: NCT01850238
Title: A 3-months Randomized, Placebo-controlled, Parallel Group, Double-blinded, Multi-centre, Phase I Study to Assess Tolerability & Safety of AADvac1 Applied to Patients With Mild-Moderate Alzheimer's Disease With 3-months Open Label Extension
Brief Title: Safety Study of AADvac1, a Tau Peptide-KLH-Conjugate Active Vaccine to Treat Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Axon Neuroscience SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AXON CO 18700; 2012-003916-29 (EudraCT Number)
Record Dates: First submitted 2013-05-07; First posted 2013-05-09 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer disease; tau protein; neurofibrillary degeneration; disease-modifying
MeSH Terms: conditions — Alzheimer Disease; Frontotemporal Dementia | interventions — AADvac1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (adjuvant in saline solution) (Placebo Comparator): Placebo patients will receive 1 dose of placebo per month over 3 months, for a total of 3 administrations.
  Placebo consists of vaccine adjuvant in saline solution. Placebo is administered subcutaneously.
  Interventions: Other: Placebo
- AADvac1 (Experimental): AADvac1 patients will receive 1 dose of AADvac1 per month over 3 months, for a total of 3 administrations.
  AADvac1 is a vaccine (single-use vials with solution ready for injection) AADvac1 is administered subcutaneously.
  Interventions: Biological: AADvac1

INTERVENTIONS:
Biological: AADvac1 — AADvac1 is intended as an active vaccination for disease-modifying treatment of Alzheimer's disease.
  Other Names: (no commercial or INN name assigned yet)
  Arms: AADvac1
Other: Placebo — The placebo contains the same buffer and adjuvant as AADvac1, but lacks the API.
  Other Names: (no other names)
  Arms: Placebo (adjuvant in saline solution)

SUMMARY:
This first-time-in-man study is mainly designed to assess the safety and tolerability of AADvac1 in the treatment of Alzheimer's disease.

AADvac1 is a vaccine directed against pathologically modified Alzheimer tau protein that is the main constituent of neurofibrillary tangles (NFTs), and is intended to be a disease-modifying treatment for Alzheimer's disease, i.e. to halt its progress.

As this study is a Phase I study focused on tolerability and safety, efficacy will be assessed in an exploratory manner.

DETAILED DESCRIPTION:
AADvac1 is a candidate therapeutic vaccine for Alzheimer's disease that targets misfolded tau protein, a common denominator of neurofibrillary pathology. Based on preclinical results, the intervention is expected to reduce the number of neurofibrillary tangles, remove hyperphosphorylated tau protein and reduce the amount of oligomerized and insoluble pathological tau in the brain, to halt the spread of neurofibrillary pathology through the brain, and thus prevent associated cognitive decline.

The vaccine's antigenic determinant is a synthetic peptide derived from a tau protein sequence, which is coupled to keyhole limpet hemocyanin (KLH) and uses aluminum hydroxide (Alhydrogel) as an adjuvant.

At present AADvac1 is intended as an active immunotherapy for patients with diagnosed Alzheimer's disease (AD). Patients will receive 3 - 6 immunization doses; the raised titers of therapeutic antibodies and possible benefits of the treatment can extend beyond the duration of the study.

Because of the central role of pathological misfolded tau protein in the etiology of AD, the vaccine is expected to be more effective than active or passive immunotherapies aiming to eliminate the amyloid β plaques that have been clinically investigated so far.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of probable Alzheimer's disease based on the NINCDS/ADRDA criteria.
2. MMSE 15-26.
3. stable dose of Alzheimer's Disease treatment since 3 months before screening visit or being untreated.
4. Hachinski Ischemia Scale ≤ 4.
5. MRI consistent with the diagnosis of AD.
6. Informed consent capability
7. Written informed consent signed and dated by the patient & caregiver.
8. Age between 50 and 85 years.
9. Availability of partner/caregiver.
10. Adequate visual and auditory abilities and German language skills for neuropsychological testing.
11. Females either surgically sterile or 2+ years postmenopausal.
12. Participant on stable doses of all medications for concomitant illnesses according to medical history for at least 30 days prior to Visit 1 if considered relevant by the investigator.
13. Sexually active males must be using reliable contraception methods or be surgically sterile.

Exclusion Criteria:

1. Pregnant women.
2. Participation in another clinical trial within 3 months before Visit 1.
3. Patients not expected to complete the clinical trial.
4. Presence or history of allergy to components of the vaccine, if considered relevant by the investigator.
5. Contraindication for MRI imaging (e.g. metallic endoprosthesis, stent implantation in the last 6 months).
6. Any of the following detected by brain MRI:

   * Thromboembolic infarction
   * Other focal lesions which may be responsible for the cognitive status of the patient
   * More than one lacunar infarct with a diameter of less than 1.5 cm in any dimension
   * Any lacunar infarct in a strategically important location such as the thalamus, hippocampus of either hemisphere, head of the left caudate
   * White matter lesions involving more than 25% of the hemispheric white matter
7. Surgery (under general anaesthesia) within 3 months prior to study entry and scheduled surgery during the whole study period.
8. History and/or presence of autoimmune disease, if considered relevant by the investigator.
9. Recent (≤3 years since last specific treatment) history of cancer (Exceptions: basal cell carcinoma, intraepithelial cervical neoplasia).
10. Active infectious disease (e.g., Hepatitis B, C).
11. Presence and/or history of Immunodeficiency (e.g., HIV).
12. Significant systemic illness, if considered relevant by the investigator.
13. Hypothyroidism (patients with corrected hypothyroidism are eligible for the study if treatment has been stable for 3 months before study entry)
14. History of significant psychiatric illness such as schizophrenia, bipolar affective disorder or major depression.
15. Current depressive episode (Geriatric Depression Scale GDS >5 at Visit 1).
16. Metabolic or toxic encephalopathy or dementia due to a general medical condition.
17. Alcoholism or substance abuse within the past year (alcohol or drug intoxication).
18. Wernicke's encephalopathy
19. History or evidence of any other CNS disorder that could be the cause of dementia (infectious or inflammatory/demyelinating CNS conditions, Creutzfeldt-Jakob disease, Parkinson's disease, Huntington's disease, brain tumour, subdural haematoma, etc.)
20. History or evidence of cerebrovascular disease (ischemic or haemorrhagic stroke, transient ischemic attack), or diagnosis of possible, probable or definite vascular dementia.
21. Epilepsy.
22. Prior and/or current treatment with experimental immunotherapeutics including IVIG or any vaccines for AD.
23. Current treatment with immunosuppressive drugs.
24. Change in dose of standard treatments for AD or hypothyroidism within 3 months prior to visit 1.
25. Change in dose of previous and current medications which the patient is taking because of consisting illnesses according medical history within the last 30 days prior to visit 1, if considered clinically relevant by the investigator.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-05; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Tolerability and safety profile of AADvac1 in patients with mild-to-moderate Alzheimer's disease | Tolerability & safety are assessed over a period of 3 months / 3 administrations
  Safety is assessed via recording of all Adverse Events and Adverse Events
  Patients are observed via:
  * MRI
  * Clinical & neuro-psychiatric observation
  * Cognitive testing
  * ECG
  * Blood biochemistry, hematology, coagulation measurement
  * Urine analysis

SECONDARY OUTCOMES:
Immunogenicity of AADvac1 | Immune response to the vaccine will be assessed over 3 months / 3 administrations
  Measurement of:
  * Titres of antibodies reactive with AADvac1
  * Titres of antibodies reactive with Alzheimer tau protein
  * Antibody isotype profiles

OTHER OUTCOMES:
Patient cognition | 3 months / 3 administrations, with an optional 3 months open label extension phase (3+3 administrations)
  Tests used:
  * ADAS-Cog (Alzheimer's Disease Assessment Scale-cognitive subscale)
  * COWAT (Controlled oral word association test)
  * Category fluency

CONTACTS AND LOCATIONS:
Overall Officials: Reinhold Schmidt, Professor, Principal Investigator — Medizinische Universität Graz
Locations (3):
- Austria (3):
  - Univeristätsklinik für Neurologie, PMU, Christian-Doppler Klinik, Salzburg, Salzburg
  - Medizinische Universitat Graz, Graz, Styria
  - Medizinische Universitat Wien, Vienna, Vienna

REFERENCES:
- [Derived] Novak P, Schmidt R, Kontsekova E, Kovacech B, Smolek T, Katina S, Fialova L, Prcina M, Parrak V, Dal-Bianco P, Brunner M, Staffen W, Rainer M, Ondrus M, Ropele S, Smisek M, Sivak R, Zilka N, Winblad B, Novak M. FUNDAMANT: an interventional 72-week phase 1 follow-up study of AADvac1, an active immunotherapy against tau protein pathology in Alzheimer's disease. Alzheimers Res Ther. 2018 Oct 24;10(1):108. doi: 10.1186/s13195-018-0436-1. PMID 30355322
- [Derived] Novak P, Schmidt R, Kontsekova E, Zilka N, Kovacech B, Skrabana R, Vince-Kazmerova Z, Katina S, Fialova L, Prcina M, Parrak V, Dal-Bianco P, Brunner M, Staffen W, Rainer M, Ondrus M, Ropele S, Smisek M, Sivak R, Winblad B, Novak M. Safety and immunogenicity of the tau vaccine AADvac1 in patients with Alzheimer's disease: a randomised, double-blind, placebo-controlled, phase 1 trial. Lancet Neurol. 2017 Feb;16(2):123-134. doi: 10.1016/S1474-4422(16)30331-3. Epub 2016 Dec 10. PMID 27955995
- [Derived] Kontsekova E, Zilka N, Kovacech B, Novak P, Novak M. First-in-man tau vaccine targeting structural determinants essential for pathological tau-tau interaction reduces tau oligomerisation and neurofibrillary degeneration in an Alzheimer's disease model. Alzheimers Res Ther. 2014 Aug 1;6(4):44. doi: 10.1186/alzrt278. eCollection 2014. PMID 25478017